CLINICAL TRIAL: NCT05726045
Title: Increasing the Smoking Cessation Success Rate by Enhancing Improvement of Self-control Through Sleep-amplified Memory Consolidation
Brief Title: Increasing Smoking Cessation Success Through Sleep-amplified Memory Consolidation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TRR265 C01-P2
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use Disorder
Keywords: Addiction; Nicotine; Smoking Cessation; Relapse; Cognitive remediation; Exercise training
MeSH Terms: conditions — Tobacco Use Disorder; Behavior, Addictive; Smoking Cessation; Recurrence | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIIT morning (Active Comparator): High-intensity interval training (HIIT) in the morning
  Interventions: Behavioral: Standard smoking cessation program (SCP)
- HIIT evening (Experimental): High-intensity interval training (HIIT) in the evening
  Interventions: Behavioral: Standard smoking cessation program (SCP); Behavioral: High-intensity interval training (HIIT evening)
- HIIT morning + CRT (Active Comparator): High-intensity interval training (HIIT) in the morning + cognitive remediation treatment (CRT)
  Interventions: Behavioral: Standard smoking cessation program (SCP); Behavioral: Cognitive remediation treatment (CRT)
- HIIT evening + CRT (Experimental): High-intensity interval training (HIIT) in the evening+ cognitive remediation treatment (CRT)
  Interventions: Behavioral: Standard smoking cessation program (SCP); Behavioral: Cognitive remediation treatment (CRT); Behavioral: High-intensity interval training (HIIT evening)

INTERVENTIONS:
Behavioral: Standard smoking cessation program (SCP) — Each subject will receive a standard SCP as group treatment once a week (1h) over six weeks. This group therapy is based on behavioural therapy and a psycho-educational approach (for more details see Batra & Buchkremer, 2004), and will be carried out by a qualified therapist.
Behavioral: Cognitive remediation treatment (CRT) — The cognitive remediation treatment (CRT) employs a chess-based battery of tasks (delivered through an app-based online tool), two times per week over six weeks (60min duration per session).
  Arms: HIIT evening + CRT; HIIT morning + CRT
Behavioral: High-intensity interval training (HIIT evening) — The high-intensity interval training will be delivered through an app environment with several choices of exercise, two times per week over six weeks.
  The training will include a 5-minutes warm-up and cool down phase. In between, participants will perform four 4-minutes blocks of exercise at high intensity, interspersed with three 3-minute blocks of low intensity (total of 35 minutes exercise).
  Arms: HIIT evening; HIIT evening + CRT

SUMMARY:
The goal of this subproject is to examine the hypothesized improvement of treatment with chess-based training and sleep enhancement, both together and on their own, in smokers.

Participants will undergo fMRI measurements, sleep monitoring. They will then be assigned to one of the four experimental groups, including high-intensity interval training with or without chess-based training.

DETAILED DESCRIPTION:
This subproject aims to improve treatment outcome in patients with tobacco use disorder (TUD) by enhancing cognitive control. Evidence from the first funding period (1st FP) indicates that enhancing cognitive control using cognitive remediation training (CRT, in our case chess-based) can improve outcomes of a standard smoking cessation program. The current project will harness three means to build on this success of enhancing cognitive control by: 1. using our tried-and-tested chess-based training, 2. improving sleep using high-intensity interval training (HIIT), 3. increasing sleep-dependent consolidation of the chess-based training (see Figure 1). We hypothesize that chess-based training and sleep enhance treatment outcome, both together and on their own. To test our hypotheses, we will combine smoking cessation treatment with the aforementioned approaches as app-based add-ons (chess-based training and HIIT). This will not only allow us to apply the training in a cost-efficient way out-side the lab, it may also increase patients' compliance.

ELIGIBILITY:
Inclusion Criteria:

* severe tobacco use disorder (TUD) according to DSM-5
* sufficient ability to communicate with investigators and answer questions in both written and verbal format
* ability to provide fully informed consent and to use self-rating scales
* right-handedness
* HIIT can be performed without the risk of side effect (medical sports check)

Exclusion Criteria:

* severe internal, neurological, and/or psychiatric comorbidities; other Axis I mental disorders other than TUD according to ICD-10 and DSM 5 (except for mild depression, i.e. F32.0, adjustment disorder and specific phobias) in the last 12 months
* history of brain injury
* severe physical diseases
* common exclusion criteria for MRI (e.g. metal, claustrophobia)
* positive drug screening (opioids, benzodiazepines, barbiturates, cocaine, amphetamines)
* psychotropic medication within the last 14 days
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Time until first severe relapse | timepoint 3: follow-up 3 months after end of SCP
  days until the first severe smoking relapse after treatment
Percentage of abstinent days | timepoint 3: follow-up 3 months after end of SCP
  Percentage of abstinent days in the 3 months after treatment
Change in smoking urges | 2 time points: before and after 6 weeks SCP
  questionnaire of smoking urges (QSU, Müller et al. 2001)
Change in neural measures of response inhibition | 2 time points: before and after 6 weeks SCP
  SST fMRI task (Gan et al., 2014)
Change in neural measures of working memory | 2 time points: before and after 6 weeks SCP
  Nback fMRI task (Charlet et al., 2014)
Change in neural functional connectivity in the salience network | 2 time points: before and after 6 weeks SCP
  resting state connectivity to seed region right anterior insula

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim; Gordon Feld, Dr., Principal Investigator — Central Institute of Mental Health, Mannheim; Karen Ersche, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Gerhardt S, Kroth M, Seeger A, Schmitt R, Fritz H, Diring L, Shevchenko Y, Ersche KD, Feld G, Vollstadt-Klein S. Increasing the smoking cessation success rate by enhancing improvement of self-control through sleep-amplified memory consolidation: protocol of a randomized controlled, functional magnetic resonance study. BMC Psychol. 2025 Feb 22;13(1):157. doi: 10.1186/s40359-025-02482-w. PMID 39987116